CLINICAL TRIAL: NCT06882525
Title: The Evaluation of the Effectiveness of Subcutaneous Lidocaine Injection in Acute Herpes Zoster Neuralgia and Post-herpetic Neuralgia
Brief Title: Subcutaneous Lidocaine Injection in Acute Herpes Zoster Neuralgia and Post-herpetic Neuralgia
Acronym: SCL-HZ/PHN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, Medical doctor, Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2-25-9924
Record Dates: First submitted 2025-03-06; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Herpes Zoster; Neuralgia, Postherpetic
Keywords: Neuralgia, Postherpetic; HERPES ZOSTER; Lidocaine
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients who are referred from the dermatology clinic or voluntarily present to our pain management (Active Comparator): The result of the study will provide insight into how much subcutaneous lidocaine injection, applied to patients with pain due to acute HZ and PHN, reduces pain, compare the effectiveness between its application in the acute and chronic phases, and determine its contribution to preventing the development of PHN. Based on the outcome, the effectiveness of this treatment can be demonstrated.
  Interventions: Procedure: Lidocaine (drug)

INTERVENTIONS:
Procedure: Lidocaine (drug) — Lidocain subcuteous infiltratyion will be done to rush area.

SUMMARY:
In this study, it was aimed to compare the effect of subcutaneous lidocaine injection, which is routinely applied in pain clinic,in patients who present with pain complaints due to acute herpes zoster and post-herpetic neuralgia, and investigate its contribution to preventing the development of post-herpetic neuralgia

DETAILED DESCRIPTION:
Herpes zoster (HZ; shingles) is a disease associated with inflammation of peripheral nerves, which can progress with acute and chronic pain, and is considered a significant cause of postherpetic neuralgia (PHN). The varicella-zoster virus (VZV) causes a primary infection known as chickenpox. The virus then migrates to spinal and cranial sensory ganglia, becoming latent through nerve axons and possibly via viremia from the skin lesions. In some individuals later in life, the virus reactivates, causing a secondary infection known as HZ. When the virus reactivates, it progresses along the affected sensory nerve, causing neuronal damage, and reaches the corresponding dermatome of the skin, leading to vesicular rashes and pain (1). There are three stages of HZ pain: the acute pain phase (up to one month), the subacute pain phase (30-90 days after lesion healing), and the PHN phase (pain lasting more than 90 days after the rash begins) (2).

Since herpes zoster can be very painful, adequate pain control is essential. The acute neuralgia of HZ typically presents as acute pain in the relevant dermatome, ranging from mild itching, tingling, and allodynia to severe pain, which often occurs before the skin lesions. For mild to moderate pain in acute HZ, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs), or tramadol can be considered. For moderate pain, opioids such as morphine or oxycodone may be administered. If moderate pain is not controlled by opioids, gabapentin or pregabalin, tricyclic antidepressants, or corticosteroids may be considered as additional treatments (3). Furthermore, in acute HZ, intradermal infiltration of local anesthetics and corticosteroids has been shown to be effective in reducing pain and preventing the development of PHN (4).

The pharmacological treatment of PHN includes a variety of medications such as alpha-2 delta ligands (gabapentin and pregabalin), other anticonvulsants (carbamazepine), tricyclic antidepressants (amitriptyline, nortriptyline), topical analgesics (5% lidocaine patch, capsaicin), tramadol, or other opioids (5). Repetitive intradermal administration of lidocaine and steroids is also used in the treatment of PHN (4).

In this study, it was aimed to demonstrate the effect of subcutaneous lidocaine injection, which is routinely administered in pain clinic, in patients presenting with pain due to acute HZ and PHN, compare its effects in the acute and chronic stages, and investigate its contribution to preventing the development of PHN. The study design and potential risks are explained in the relevant sections.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18
* with acute HZ pain (rash duration < 30 days
* pain due to PHN (rash duration > 3 months),

Exclusion Criteria:

patients on anticoagulants or have coagulation disorders, patients with psychomotor disorders patients with uncontrolled diabetes patients with bacterial infection or infectious discharge in the affected dermatomal region patients allergic to lidocaine patients with lesions in the facial or genital regions pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-07 (Estimated); Primary Completion 2025-09-07 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
NRS , DN4 | 1st week after injection
  The patients' pain scores will be assessed before treatment using the NRS (Numerical Rating Scale) and DN4 (Douleur Neuropathique en 4 Questions) pain scales. During the treatment process, patients will receive three injections, one week apart, and the NRS and DN4 pain scores will be reassessed one week after each injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Üniversiteler Mahallesi 1604. Cadde No: 9 Çankaya/ANKARA, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Privacy.

REFERENCES:
- [Background] Johnson RW, Alvarez-Pasquin MJ, Bijl M, Franco E, Gaillat J, Clara JG, Labetoulle M, Michel JP, Naldi L, Sanmarti LS, Weinke T. Herpes zoster epidemiology, management, and disease and economic burden in Europe: a multidisciplinary perspective. Ther Adv Vaccines. 2015 Jul;3(4):109-20. doi: 10.1177/2051013615599151. PMID 26478818